CLINICAL TRIAL: NCT05283889
Title: The Safety and Efficacy of Genicular Radiofrequency Ablation for Patients With Persistent Knee Pain Following Total Knee Arthroplasty - A Triple Blinded Randomized Sham-Controlled Trial
Brief Title: Genicular Radiofrequency Ablation Following Total Knee Arthroplasty
Acronym: GRATKA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: REB21-2105
Record Dates: First submitted 2022-02-18; First posted 2022-03-17 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Osteoarthritis, Knee
Keywords: Genicular Radiofrequency Ablation; Randomized Controlled Trial; Knee Pain; Balance
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Triple blinding will be accomplished as follows: operator (RF generator operated by assistant out of sight of operator); participant (local anesthetic administration and cannula placement identical; RF generator makes the same beeping sound for the same duration); assessor (only the study coordinator is aware of group assignment).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (GRFA) (Experimental): After the cannulae are placed and tines deployed, a single lesion (30 second ramp-up time; 80C x 2 minutes) will be made at each of the medial and lateral branches of the nerve to the vastus intermedialis, nerves to the vastus lateralis and medialis, recurrent fibular nerve, inferior medial genicular nerve. One bipolar strip lesion (intercannula distance 1.5 cm; anticipated strip lesion length 2.0 cm) at the superior medial and lateral genicular nerves will be made to accommodate anatomical variability.
  Interventions: Procedure: Genicular Radiofrequency Ablation
- Group 2 (Sham) (Active Comparator): The same procedure will be employed as per Group 1 - However, the sham procedure will involve no electrical signal applied to the participant.
  Interventions: Procedure: Sham Genicular Radiofrequency Ablation

INTERVENTIONS:
Procedure: Genicular Radiofrequency Ablation — After the cannulae are placed and tines deployed, a single lesion (30 second ramp-up time; 80C x 2 minutes) will be made at each of the medial and lateral branches of the nerve to the vastus intermedialis, nerves to the vastus lateralis and medialis, recurrent fibular nerve, inferior medial genicular nerve. One bipolar strip lesion (intercannula distance 1.5 cm; anticipated strip lesion length 2.0 cm) at the superior medial and lateral genicular nerves will be made to accommodate anatomical variability.
  Arms: Group 1 (GRFA)
Procedure: Sham Genicular Radiofrequency Ablation — After the cannulae are placed and tines deployed, a single lesion (no electrical signal applied to patient) will be made at each of the medial and lateral branches of the nerve to the vastus intermedialis, nerves to the vastus lateralis and medialis, recurrent fibular nerve, inferior medial genicular nerve. One bipolar strip lesion (intercannula distance 1.5 cm; anticipated strip lesion length 2.0 cm) at the superior medial and lateral genicular nerves will be made to accommodate anatomical variability.
  Arms: Group 2 (Sham)

SUMMARY:
Currently, nearly 1 million total knee arthroplasties (TKA) are performed yearly in the United States. Three million are projected to be performed in 2040. Between 15-30% of all patients who undergo TKA have continued pain, reduced quality of life and functional impairments that cannot be attributed to hardware failure/loosening or infection. Treatment options for persistent post TKA pain (failed TKA) are limited. There is a need for minimally invasive, and effective pain and disability modulating interventions for patients with failed TKA. Genicular radiofrequency ablation (GRFA) has been described, refined, and validated as an effective minimally invasive intervention to control refractory knee pain secondary to knee osteoarthritis (OA) as evidenced by three favorable meta-analyses published in 2021 alone.3-5 GRFA is a minimally invasive percutaneous procedure that utilizes thermal energy to coagulate nerves from the knee. Though sometimes used in practice, there is limited research describing and evaluating GRFA for patients with failed TKA. This will be the first trial to evaluate the safety and efficacy of GRFA in patients with failed TKA using a robust study design and up-to-date, evidence-based selection criteria and technique.

DETAILED DESCRIPTION:
The general objective of this study is to determine the safety and efficacy of GRFA in patients with failed TKA. The central hypothesis is that GRFA is safe and more efficacious in improving pain and function than sham GRFA. A triple blinded randomized sham-controlled trial design will be used. Patients with failed TKA will be recruited and randomized into either a thermal or sham GRFA group. Patient selection criteria and GRFA procedural technique will incorporate refinements based on expanded understanding from recent research. Outcomes will be assessed prior to and at 3, 6 and 12 months post-GRFA. The primary outcome measures will be between group difference in the change in pain (NRS) between pre- and 6 months post. Secondary outcomes will include safety and changes in function (WOMAC; sit-stand test; strength; range of motion & balance), participants' impression of change, perceived need for revision arthroplasty, analgesic use, and quality-of-life. Crossover will be offered to participants in the sham group at 6 months post-treatment. Data will be analyzed using descriptive, linear mixed-effects model and Kaplan-Meier Survival Curve statistics. The proposed research is innovative and important as it uses a robust study design to evaluate the safety and efficacy of an emerging RFA intervention in a prevalent suffering patient population.

ELIGIBILITY:
Inclusion Criteria:

* >1 year post TKA
* persistent knee pain > 4/10 in intensity on average over the prior week of one of the post-TKA knees
* refractory to conventional treatment (i.e., physiotherapy, medication, etc.)
* ≥80% pain relief with a single fluoroscopically guided local anesthetic block using 0.5 mL of 2% lidocaine for the medial and lateral branches of the nerve to the vastus intermedialis, nerve to the vastus lateralis*, inferior medial genicular nerve, infrapatellar branch of the saphenous nerve, and the recurrent fibular nerve. 0.5 mL will be injected over 2 spots (1.5 cm apart) for each of the superior medial and lateral genicular nerves corresponding to the sites of the RF cannulae for the bipolar strip lesions. *Blocks will be combined fluoroscopy/ultrasound guided.

Exclusion Criteria:

* Infection (peri-prosthetic, joint, systemic, skin/soft tissue overlying the knee to be treated)
* Prosthetic loosening or failure, periprosthetic fracture
* Severe psychiatric disorder
* Non-genicular lower extremity pain source from the spine (i.e., radiculopathy or neurogenic claudication) or peripheral joints (i.e., hip osteoarthritis)
* Peripheral vascular disease causing vascular claudication
* Connective tissue/inflammatory joint disease/widespread soft tissue pain disorder
* Poor tolerance of injection procedures (as observed from the prognostic local anesthetic blocks)
* Allergy to local anesthetic, synovial expansion into the anticipated path(s) of the local anesthetic needle/RF cannula as determined by ultrasound scanning
* Uncontrolled bleeding diathesis
* Pregnancy
* Pacemaker or neurostimulator
* Inability to complete Patient-Reported Outcome Measures due to cognitive or language limitations.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-05-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Average Pain Intensity Over the Prior week (0 - 10) | 6 months
  Numerical pain rating scale (0 - 10) with higher scores indicating a worse outcome
Change in pain intensity between pre- and 6-months post-intervention | 6 months
  Numerical Pain rating scale (NPRS) 6 month minus NPRS pre-intervention, with increased negative scores indicating a better outcome

SECONDARY OUTCOMES:
Average Pain Intensity Over the Prior Week (0 - 10) | 3 and 12-months post-intervention
  Numerical pain rating scale (0 - 10) with higher scores indicating worse outcomes
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | 3, 6 and 12-months post-intervention
  Measure of pain (0 - 20), stiffness (0 - 8) and physical function (0 - 68) with higher scores indicating wore pain, stiffness and functional limitations
The Clinical Global Impressions Scale (CGI) | 3, 6 and 12-months post-intervention
  Patient reported global impression of change (1 = Very Much Improved to 7 = Very Much Worse)
Safety - Adverse Events | 1-week, 3, 6 and 12-months post-intervention
  Presence of self-reported complications
Proportion of participants exceeding 50% pain relief | 6 months
  Proportion of participants that experience ≥ 50% pain relief
Proportion of participants exceeding Minimal Clinically Important Difference (MCID) pain relief | 6 months
  Proportion of participants that experience MCID knee pain relief
Perceived Need for Revision Arthroplasty | Baseline (Prior to), 3, 6 and 12-months post-intervention
  "If revision surgery of your knee replacement was available to you, how interested would you be in having it at this time?" Y or N
Analgesic Use | Baseline (Prior to), 3, 6 and 12-months post-intervention
  Quantitative Analgesic Questionnaire
Health-related Quality of Life | Baseline (Prior to), 3, 6 and 12-months post-intervention
  EQ-5D-5L

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Smith, PhD, Principal Investigator — University of Calgary
Locations (1):
- Vivo Cura Health, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singh JA, Yu S, Chen L, Cleveland JD. Rates of Total Joint Replacement in the United States: Future Projections to 2020-2040 Using the National Inpatient Sample. J Rheumatol. 2019 Sep;46(9):1134-1140. doi: 10.3899/jrheum.170990. Epub 2019 Apr 15. PMID 30988126
- [Background] Beswick AD, Wylde V, Gooberman-Hill R, Blom A, Dieppe P. What proportion of patients report long-term pain after total hip or knee replacement for osteoarthritis? A systematic review of prospective studies in unselected patients. BMJ Open. 2012 Feb 22;2(1):e000435. doi: 10.1136/bmjopen-2011-000435. Print 2012. PMID 22357571
- [Background] Zhang H, Wang B, He J, Du Z. Efficacy and safety of radiofrequency ablation for treatment of knee osteoarthritis: a meta-analysis of randomized controlled trials. J Int Med Res. 2021 Apr;49(4):3000605211006647. doi: 10.1177/03000605211006647. PMID 33887985
- [Background] Li G, Zhang Y, Tian L, Pan J. Radiofrequency ablation reduces pain for knee osteoarthritis: A meta-analysis of randomized controlled trials. Int J Surg. 2021 Jul;91:105951. doi: 10.1016/j.ijsu.2021.105951. Epub 2021 Apr 18. PMID 33882358
- [Background] Chen AF, Mullen K, Casambre F, Visvabharathy V, Brown GA. Thermal Nerve Radiofrequency Ablation for the Nonsurgical Treatment of Knee Osteoarthritis: A Systematic Literature Review. J Am Acad Orthop Surg. 2021 May 1;29(9):387-396. doi: 10.5435/JAAOS-D-20-00522. PMID 32701684
- [Background] Protzman NM, Gyi J, Malhotra AD, Kooch JE. Examining the feasibility of radiofrequency treatment for chronic knee pain after total knee arthroplasty. PM R. 2014 Apr;6(4):373-6. doi: 10.1016/j.pmrj.2013.10.003. Epub 2013 Dec 27. PMID 24373908
- [Background] Kapural L, Lee N, Neal K, Burchell M. Long-Term Retrospective Assessment of Clinical Efficacy of Radiofrequency Ablation of the Knee Using a Cooled Radiofrequency System. Pain Physician. 2019 Sep;22(5):489-494. PMID 31561648
- [Background] Koshi E, Cheney CW, Sperry BP, Conger A, McCormick ZL. Genicular Nerve Radiofrequency Ablation for Chronic Knee Pain Using a Three-Tined Electrode: A Technical Description and Case Series. Pain Med. 2020 Dec 25;21(12):3344-3349. doi: 10.1093/pm/pnaa204. PMID 32984887
- [Background] Erdem Y, Sir E. The Efficacy of Ultrasound-Guided Pulsed Radiofrequency of Genicular Nerves in the Treatment of Chronic Knee Pain Due to Severe Degenerative Disease or Previous Total Knee Arthroplasty. Med Sci Monit. 2019 Mar 12;25:1857-1863. doi: 10.12659/MSM.915359. PMID 30858350
- [Background] Qudsi-Sinclair S, Borras-Rubio E, Abellan-Guillen JF, Padilla Del Rey ML, Ruiz-Merino G. A Comparison of Genicular Nerve Treatment Using Either Radiofrequency or Analgesic Block with Corticosteroid for Pain after a Total Knee Arthroplasty: A Double-Blind, Randomized Clinical Study. Pain Pract. 2017 Jun;17(5):578-588. doi: 10.1111/papr.12481. Epub 2016 Sep 19. PMID 27641918
- [Background] Fonkoue L, Steyaert A, Kouame JK, Bandolo E, Lebleu J, Fossoh H, Behets C, Detrembleur C, Cornu O. A Comparison of Genicular Nerve Blockade With Corticosteroids Using Either Classical Anatomical Targets vs Revised Targets for Pain and Function in Knee Osteoarthritis: A Double-Blind, Randomized Controlled Trial. Pain Med. 2021 May 21;22(5):1116-1126. doi: 10.1093/pm/pnab014. PMID 33772285
- [Background] Tran J, Peng PWH, Lam K, Baig E, Agur AMR, Gofeld M. Anatomical Study of the Innervation of Anterior Knee Joint Capsule: Implication for Image-Guided Intervention. Reg Anesth Pain Med. 2018 May;43(4):407-414. doi: 10.1097/AAP.0000000000000778. PMID 29557887
- [Background] Cushman DM, Monson N, Conger A, Kendall RW, Henrie AM, McCormick ZL. Use of 0.5 mL and 1.0 mL of Local Anesthetic for Genicular Nerve Blocks. Pain Med. 2019 May 1;20(5):1049-1052. doi: 10.1093/pm/pny277. No abstract available. PMID 30590798
- [Background] Roos EM, Klassbo M, Lohmander LS. WOMAC osteoarthritis index. Reliability, validity, and responsiveness in patients with arthroscopically assessed osteoarthritis. Western Ontario and MacMaster Universities. Scand J Rheumatol. 1999;28(4):210-5. doi: 10.1080/03009749950155562. PMID 10503556
- [Background] Kreibich DN, Vaz M, Bourne RB, Rorabeck CH, Kim P, Hardie R, Kramer J, Kirkley A. What is the best way of assessing outcome after total knee replacement? Clin Orthop Relat Res. 1996 Oct;(331):221-5. doi: 10.1097/00003086-199610000-00031. PMID 8895642
- [Background] Grafton ST, Ralston AB, Ralston JD. Monitoring of postural sway with a head-mounted wearable device: effects of gender, participant state, and concussion. Med Devices (Auckl). 2019 May 1;12:151-164. doi: 10.2147/MDER.S205357. eCollection 2019. PMID 31118838
- [Background] Busner J, Targum SD. The clinical global impressions scale: applying a research tool in clinical practice. Psychiatry (Edgmont). 2007 Jul;4(7):28-37. PMID 20526405
- [Background] Robinson-Papp J, George MC, Wongmek A, Nmashie A, Merlin JS, Ali Y, Epstein L, Green M, Serban S, Sheth P, Simpson DM. The Quantitative Analgesic Questionnaire: A Tool to Capture Patient-Reported Chronic Pain Medication Use. J Pain Symptom Manage. 2015 Sep;50(3):381-6. doi: 10.1016/j.jpainsymman.2015.03.013. Epub 2015 Apr 23. PMID 25912277
- [Background] Balestroni G, Bertolotti G. [EuroQol-5D (EQ-5D): an instrument for measuring quality of life]. Monaldi Arch Chest Dis. 2012 Sep;78(3):155-9. doi: 10.4081/monaldi.2012.121. Italian. PMID 23614330
- [Background] Kim SY, Le PU, Kosharskyy B, Kaye AD, Shaparin N, Downie SA. Is Genicular Nerve Radiofrequency Ablation Safe? A Literature Review and Anatomical Study. Pain Physician. 2016 Jul;19(5):E697-705. PMID 27389113